CLINICAL TRIAL: NCT02346981
Title: Chronic Resistance Training and Post-exercise Blood Pressure in Normotensive Older Women
Brief Title: Resistance Training and Post-exercise Blood Pressure in Normotensive Older Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Estadual de Londrina (Other)
Responsible Party: Principal Investigator, Aline Mendes Gerage, Master student, Universidade Estadual de Londrina
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PIUEL2008
Record Dates: First submitted 2015-01-20; First posted 2015-01-27 (Estimated); Last update posted 2015-01-28 (Estimated); Status verified 2015-01

CONDITIONS: Healthy Older Adults
MeSH Terms: interventions — Resistance Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention gruop (Experimental): The intervention group was submitted to a resistance training program that consisted of eight exercises performed in two sets of 10 to 15 repetitions, three times per week.
  Interventions: Behavioral: Resistance training
- Control group (No Intervention): The control group performed a stretching training program for the major muscle groups, in sessions of 30 minutes, twice a week

INTERVENTIONS:
Behavioral: Resistance training — Supervised resistance training program was performed on three nonconsecutive days per week at morning period for 12 weeks. The resistance training program included eight exercises in two consecutive sets of 10-15 repetitions until moderate fatigue, except for crunch exercise which was performed on 20 to 30 repetitions without overload. The participants were instructed to perform repetitions at a ratio of 1:2 (concentric and eccentric phases, respectively). Subjects rested for 60- to 90-s between each set and for 2- to 3-min between each exercise. Each subject was individually supervised. Increases of 2-5 % for the upper limb exercises and 5-10 % for the lower limb exercises every time that subjects were able to complete 15 repetitions in both sets.
  Arms: Intervention gruop

SUMMARY:
The purpose of the present study was to analyze the effect of 12 weeks of resistance training on post-exercise blood pressure (BP) and to to correlate the acute and chronic decrease in blood pressure (BP) following resistance training in normotensive older women. Twenty-eight older women were randomly assigned to a training group (TG) or to a control group (CG). The TG underwent a resistance training program (8 exercises, 2 sets, 10-15 repetitions), while the CG performed stretching exercises (2 sets, 20 s each, 2 nonconsecutive days/week). Both groups performed the intervention for 12 weeks. At baseline and after intervention the subjects were submitted to two sessions: resistance exercise session and control session. In these sessions, BP was obtained in pre and post-sessions. Rest blood pressure were also measure at baseline and after 12 weeks of intervention.

DETAILED DESCRIPTION:
Older (≥60 years) normotensive and physically inactive women were recruited. Women were randomized into training group (TG) or control group (CG) and submitted to 12 weeks of intervention. The intervention programs were divided into three phases: initial (first two weeks), intermediate (from week 3 to week 10) and final (last two weeks). The TG was submitted to a resistance training program that consisted of eight exercises performed in two sets of 10 to 15 repetitions, three times per week. The CG performed a stretching training program for the major muscle groups, in sessions of 30 minutes, twice a week. These interventions were maintained during the 12 weeks.

During initial and final phases subjects of both groups were submitted to two acute experimental sessions: resistance exercise and control, which were performed in random order. The resistance exercise session was similar to those performed during the resistance training program (i.e., 7 exercises, 2 sets, 10-15 repetitions). In the control session participants remained seated for 40 min. Before and after each session the BP parameters were obtained. The chronic effect of resistance training on post-exercise BP were assessed by analyzing the changes (∆) in BP after acute experimental sessions at initial and final phases. The correlation between acute and chronic responses of blood pressure following resistance training was analyses correlating the acute blood pressure observed in initial phase with the chronic effect of resistance training on rest blood pressure.

ELIGIBILITY:
Inclusion Criteria:

* normotensive female;
* aged 60-to-80 years old;
* nonsmokers;
* without diabetes, cardiac disease or renal dysfunction;
* not practicing regular physical activity over the six months preceding the beginning of the investigation;
* being free of any musculoskeletal or other disorders that might affect their ability to participate in the study,
* should not be taking drugs with inotropic or chronotropic actions;
* should not be using hormonal replacement therapy;
* have no restriction for participation in physical exercise, after diagnostic, graded exercise stress test with 12-lead ECG.

Exclusion Criteria:

* insufficient attendance to the training sessions (< 85 % of the total sessions);
* unavailability of time to perform the evaluations

Ages: 60 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2008-02; Primary Completion 2008-06 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
changes in clinic blood pressure | baseline, 12 weeks

SECONDARY OUTCOMES:
changes in post-exercise blood pressure | baseline, 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Aline M Gerage, Master, Principal Investigator — Universidade Estadual de Londrina; Edilson S Cyrino, Doctor, Study Director — Universidade Estadual de Londrina

REFERENCES:
- [Derived] Gerage AM, Ritti-Dias RM, do Nascimento MA, Pina FL, Goncalves CG, Sardinha LB, Cyrino ES. Chronic resistance training does not affect post-exercise blood pressure in normotensive older women: a randomized controlled trial. Age (Dordr). 2015 Jun;37(3):63. doi: 10.1007/s11357-015-9801-1. Epub 2015 Jun 6. PMID 26047957